CLINICAL TRIAL: NCT00940732
Title: The Elite Athlete Mental Health Strategy: A Randomised Controlled Trial of an Online Intervention for the Mental Health Help-Seeking of Elite Athletes
Brief Title: The Elite Athlete Mental Health Strategy Trial
Acronym: TEAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amelia Gulliver (Other)
Collaborators: Australian Institute of Sport (Other)
Responsible Party: Sponsor-Investigator, Amelia Gulliver, Ms Amelia Gulliver, Australian National University
Organization: Australian National University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2009/373
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Mental Health Help-Seeking
Keywords: Help-seeking; Mental Health; Athletes
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Destigmatisation and Mental Health Literacy (Experimental)
  Interventions: Other: Destigmatisation and Mental Health Literacy
- Help-seeking list (Experimental)
  Interventions: Other: Help-seeking list
- Feedback (Experimental)
  Interventions: Other: Feedback
- Control (No Intervention)

INTERVENTIONS:
Other: Destigmatisation and Mental Health Literacy — Written material delivered over 2 weeks via the Internet, including "mythbusters", debunking common myths around anxiety and depression, as well information about a range of celebrities who have identified themselves as having depression or anxiety. Also contains mental health literacy information.
  Arms: Destigmatisation and Mental Health Literacy
Other: Help-seeking list — List of sources for mental health help-seeking delivered over 2 weeks.
  Arms: Help-seeking list
Other: Feedback — Written material delivered over 2 weeks via the Internet, including two short self-report measures (Goldberg Anxiety, Goldberg Depression), which will provide feedback to the participant about levels of depression and anxiety.
  Arms: Feedback

SUMMARY:
The purpose of this study is to determine whether positive mental health help-seeking attitudes, and behaviour in elite athletes can be increased through an online intervention.

DETAILED DESCRIPTION:
Mental disorders account for approximately 30% of the non-fatal disease burden in Australia, with the most prevalent disorders of depression, anxiety and substance use disorders experienced by 18% of the population in any single year. These disorders are significantly more common in young adulthood than at any other stage in the lifespan. Despite the availability of effective treatments for many disorders, this high susceptibility in young people is coupled with low rates of seeking professional help. As elite athletes have been found to have less positive attitudes towards seeking help for mental health issues, and they are most often young adults themselves, they may be even less likely than non-athletes to utilise professional services. Although there is a strong relationship between exercise and positive mental health, the prevalence of mental disorders in elite athletes is currently not known. A literature review of the general literature on help seeking and a series of focus groups with elite athletes from the Australian Institute of Sport conducted by the current research group in 2008, suggested that help-seeking by these athletes might be increased by improving their knowledge about mental health, reducing stigma, and providing feedback about the symptoms of common mental disorders.

The current project was designed to test these possibilities utilising an online format. The Elite Athlete Mental health Strategy (TEAMS) project comprises two phases: (1) a large scale survey of the mental health status of elite athletes; (2) a randomised controlled trial of the effectiveness of three interventions designed to increase help seeking attitudes and help seeking behaviours related to mental disorders in elite athletes. These three interventions are: destigmatisation and mental health literacy; feedback; and a help-seeking list of resources. The study aims to compare the effectiveness of these three interventions relative to each other and a control condition.

ELIGIBILITY:
Inclusion Criteria:

* Invited through sports organisation
* Elite athlete
* Able to read English

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Help-seeking attitudes (Attitudes Toward Seeking Professional Psychological Help: Shortened Form, ATSPPH-SF) | Baseline, post, 3 month, and 6 month follow-up

SECONDARY OUTCOMES:
Help-seeking behaviour, and Help-seeking intentions (General Help-Seeking Questionnaire, GHSQ) | Baseline, post, 3 month, and 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Gulliver, BA, BAppPsych, BScPsych (Hons), Principal Investigator — The Centre for Mental Health Research, The Australian National University; Kathy Griffiths, BSc (Hons), PhD, Study Chair — The Centre for Mental Health Research, The Australian National University; Helen Christensen, BA (Hons), MPsych, PhD, Study Director — The Centre for Mental Health Research, The Australian National University
Locations (1):
- The Centre for Mental Health Research, The Australian National University, Canberra, Australian Capital Territory, Australia

REFERENCES:
- [Derived] Gulliver A, Griffiths KM, Christensen H, Mackinnon A, Calear AL, Parsons A, Bennett K, Batterham PJ, Stanimirovic R. Internet-based interventions to promote mental health help-seeking in elite athletes: an exploratory randomized controlled trial. J Med Internet Res. 2012 Jun 29;14(3):e69. doi: 10.2196/jmir.1864. PMID 22743352